CLINICAL TRIAL: NCT06797843
Title: Clinical Evaluation of Bioactive Resin Composites Versus Caries Control Technique in Management of Class I Carious Cavities in High Caries Risk Patients: a Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mansour Khalil Mansour, Dr. Sara Mansour Khalil, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14422023456853
Record Dates: First submitted 2025-01-21; First posted 2025-01-29 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: High Caries Risk Patients
Keywords: high caries risk patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- "SPRG-based" Resin Composite. (BEAUTIFIL II, Shofu Inc. Kyoto, Japan). (Experimental): A fluoride releasing, highly aesthetic dental material for all classes of restorations with S-PRG (Surface Pre-reacted Glass Ionomer) technology in regards to it's ability to recharge fluoride and appropriate for patients with a high caries index.
  Interventions: Other: "SPRG-based" Resin Composite : (BEAUTIFIL II, Shofu Inc. Kyoto, Japan).
- "Alkasite-based" restoration. (Cention N) (Experimental): Cention N offers tooth-coloured esthetics together with high flexural strength. The new filling material belongs to the materials group of Alkasites. The patented alkaline filler increases the release of hydroxide ions to regulate the pH value during acid attacks. As a result, demineralization can be prevented. Moreover, the release of large numbers of fluoride and calcium ions forms a sound basis for the remineralization of dental enamel. The initiator system enables good chemical self-curing.
- Provisional RMGI(Fuji IX EXTRA),followed by nanohybrid resin composite(Neo Spectra® ST LV, Dentsply) (Active Comparator): Traditional caries control technique by provisional Resin Modified Glass ionomer for 3 months period and then followed by removal and application of conventional nano hybrid composites.
  Interventions: Other: provisional Resin modified glass ionomer followed by Nanohybrid composite

INTERVENTIONS:
Other: "SPRG-based" Resin Composite : (BEAUTIFIL II, Shofu Inc. Kyoto, Japan). — A fluoride releasing, highly aesthetic dental material that is S-PRG (Surface Pre-reacted Glass Ionomer) based , has the ability to recharge fluoride and appropriate for patients with a high caries index.
  Arms: "SPRG-based" Resin Composite. (BEAUTIFIL II, Shofu Inc. Kyoto, Japan).
Other: Alkasite based restoration : Cention N — Cention N offers tooth-coloured esthetics together with high flexural strength. The new filling material belongs to the materials group of Alkasites. The patented alkaline filler increases the release of hydroxide ions to regulate the pH value during acid attacks. As a result, demineralization can be prevented. Moreover, the release of large numbers of fluoride and calcium ions forms a sound basis for the remineralization of dental enamel. The initiator system enables good chemical self-curing.
Other: provisional Resin modified glass ionomer followed by Nanohybrid composite — GC Fuji IX GP® EXTRA is the fastest setting glass ionomer on the market.The faster final set saves valuable chair time which provides improved stability against water, an important feature in challenging oral environments. This product contains a next generation glass filler which elicits higher translucency, fluoride release, reactivity and a faster setting time.
  Then followed by Conventional Nano hybrid composite restoration(Neo Spectra® ST LV, Dentsply Sirona) which is nano-ceramic, light-cured, radiopaque, universal composite with novel SphereTEC filler technology.
  Other Names: Traditional Caries Control Technique
  Arms: Provisional RMGI(Fuji IX EXTRA),followed by nanohybrid resin composite(Neo Spectra® ST LV, Dentsply)

SUMMARY:
The aim of the study is to clinically evaluate the performance of S-PRG based & Alkasite based resin composite restorations versus conventional resin composite restorations after caries control in Class I carious cavities in posterior molar teeth over 1 year follow up.

DETAILED DESCRIPTION:
Traditionally, less conservative methods have been employed to treat tooth decay, which implied more loss of healthy dental tissue in order to increase the mechanical retention of the restorative material. Minimally invasive treatments have been proposed as an alternative therapy, which has evolved in with the development of new biomaterials.Bioactive restorative materials, as advocated by the FDI World Dental Federation, can promote mineralization/hard tissue creation, bacterial infection control, inflammation prevention, and tissue regeneration. In simpler terms : One efficient way to achieve bioactive functionalities in dental materials is to use particles that have the ability to release particular component.The development of "Giomer" based resin composites, which have the added benefit of prolonged fluoride and other ions release as well as rechargeability, is one of the key technological advances in resin composites to promote its usage as a bioactive material.In fact, Giomers with S-PRG fillers can release more fluoride than that of other fluoride-releasing restorations.Acid neutralization capacity by S-PRG fillers, one of many bioactive functions, is in which the pH of the surrounding environment became slightly alkaline upon contact with water or acidic solutions, exhibiting a modulation impact on acidic circumstances. Owing to the release of multiple ions, such modulation effect might be brought about by the release of Sr, B, Na, and F ions clarifying an acid buffering mechanism.A modification of GIC is Cention-N, which was introduced as a new resin-based material containing alkacid fillers, such as fluoride, calcium, and hydroxide ions, to neutralize acids. Owing to being tooth-colored, inexpensive, and having good flexural strength, It's considered as a subcategory of the composite material class.With properties similar to those of GICs and RBCs, Cention-N releases calcium, hydroxyl, and fluoride ions to prevent tooth demineralization. The presence of hydroxide ions on the material's surface may be crucial in neutralizing the acids that were produced by cariogenic bacteria Additionally, the filler's release of calcium and fluoride ions contributes in remineralization process.In Conclusion; S-PRG & Alkasite based composite restorative materials are able to release ions that contribute to tooth mineralization as well as have a modulation effect on the acidic conditions produced by oral cariogenic microorganisms.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion:

  1. Adult Patients (Male or Females) aging ≥21-50 years.
  2. Patients with high level of caries risk.
  3. Patients with good likelihood of recall availability.

Tooth inclusion:

1- Permanent posterior molar teeth with primary simple occlusal Class I carious lesions (ICDAS 3 or 4 scores) 3- 2- Vital, periodontally sound and with positive reaction to cold stimulus. 4- 3-Well-formed and fully erupted in normal functional occlusion with natural antagonist and adjacent teeth

Exclusion Criteria:

- Participants with general/systemic illness. 2- Pregnant or lactating females. 3- Concomitant participation in another research study. 4- Inability to comply with study procedures. 5- Heavy bruxism habits. 6- Last experience with allergic reactions against any components of the used materials.

7- Patients receiving orthodontic treatment.

Tooth exclusion:

1. Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
2. Non-vital teeth, Fractured or cracked teeth.
3. Secondary carious lesions.
4. Hypocalcified or hypoplastic teeth.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative (hypersensitivity) and tooth vitality. | at baseline, 3 months, 6 months and 12 months.
  Revised FDI Criteria for Biological properties and by scoring:
  1. clinically very good
  2. clinically good
  3. clinically sufficient
  4. clinically unsatisfactory
  5. clinically poor
Caries at restoration margin (CAR). | at baseline,3 months, 6 months and 12 months.
  Revised FDI Criteria for Biological properties and by scoring:
  1. clinically very good
  2. clinically good
  3. clinically sufficient
  4. clinically unsatisfactory
  5. clinically poor

SECONDARY OUTCOMES:
Cost effectiveness | at baseline, 3 months, 6 months and 12 months.
  A. Cost of single restoration at baseline (for both groups) (Mean, ±SD). B. Average cost per restoration after1 year (Mean, ±SD).
  * - (for intervention group in case of adverse effects) (Mean, ±SD).
  * - (for control group: cost of the replacement with final restoration) in addition to the cost of adverse effects (Mean, ±SD).